CLINICAL TRIAL: NCT00284713
Title: Transplantation Of Progenitor Cells And Recovery Of Left Ventricular Function In Patients With Nonischemic Dilatative Cardiomyopathy
Brief Title: Progenitor Cell Therapy in Dilative Cardiomyopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPCARE-DCM
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Heart Failure, Congestive; Cardiomyopathy, Dilated; Stem Cell Transplantation
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: intracoronary infusion of BMC — catheter delivery of stem cells

SUMMARY:
Intracoronary infusion of bone marrow derived progenitor cells into the LAD in patients with non ischemic dilated cardiomyopathy.

DETAILED DESCRIPTION:
Initial clinical pilot trials suggested that intracoronary infusion of bone marrow-derived progenitor cells (BMC) may enhance left ventricular functional recovery in patients with acute myocardial infarction. It is unknown, however, whether such a strategy might also be applicable to patients with non-ischemic dilated cardiomyopathy (DCM). Therefore, we initiated the TOPCARE-DCM - trial (Transplantation Of Progenitor Cells And Recovery of Left Ventricular Function in Patients with non ischemic Dilatative CardioMyopathy) aiming to regionally improve left ventricular contractility by selective infusion of BMC into the left anterior descending coronary artery.

Patients will be randomized 2:1 (20/10) BMC Infusion versus standard medical therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 8-80
* Dilated Cardiomyopathy, Ejection fraction < 40%
* LVEDD > 60mm
* Stable clinical condition within last 6 months
* Written informed consent

Exclusion Criteria:

* Myocardial infarction or coronary intervention in the past
* Change of medical therapy within the last 6 weeks prior to cell therapy
* Tumor within last 5 years or incomplete remission
* Active infection
* Active bleeding
* Stroke within last 2 years
* Surgery or trauma within last 2 months
* Uncontrolled hypertension
* HIV infection
* Chronic inflammatory disease
* Liver disease (GOT > 2x upper normal limit)
* Renal dysfunction (creatinin > 2.0mg/dl)
* Thrombopenia < 100.000
* Anemia (hemoglobin < 8.5 g/dl)
* Mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
LV function (Ejection fraction within 3 months) Simpson | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, Principal Investigator — Div. of Cardiology, University of Frankfurt, Germany

REFERENCES:
- [Derived] De Rosa S, Seeger FH, Honold J, Fischer-Rasokat U, Lehmann R, Fichtlscherer S, Schachinger V, Dimmeler S, Zeiher AM, Assmus B. Procedural safety and predictors of acute outcome of intracoronary administration of progenitor cells in 775 consecutive procedures performed for acute myocardial infarction or chronic heart failure. Circ Cardiovasc Interv. 2013 Feb;6(1):44-51. doi: 10.1161/CIRCINTERVENTIONS.112.971705. Epub 2013 Jan 29. PMID 23362308
- [Derived] Leistner DM, Seeger FH, Fischer A, Roxe T, Klotsche J, Iekushi K, Seeger T, Assmus B, Honold J, Karakas M, Badenhoop K, Frantz S, Dimmeler S, Zeiher AM. Elevated levels of the mediator of catabolic bone remodeling RANKL in the bone marrow environment link chronic heart failure with osteoporosis. Circ Heart Fail. 2012 Nov;5(6):769-77. doi: 10.1161/CIRCHEARTFAILURE.111.966093. Epub 2012 Aug 30. PMID 22936827
- [Derived] Xu Q, Seeger FH, Castillo J, Iekushi K, Boon RA, Farcas R, Manavski Y, Li YG, Assmus B, Zeiher AM, Dimmeler S. Micro-RNA-34a contributes to the impaired function of bone marrow-derived mononuclear cells from patients with cardiovascular disease. J Am Coll Cardiol. 2012 Jun 5;59(23):2107-17. doi: 10.1016/j.jacc.2012.02.033. PMID 22651868